CLINICAL TRIAL: NCT03994809
Title: International Cross-sectional Study on the Effectiveness of Biofield Therapy for the Relief of Various Symptoms
Brief Title: International Study of Biofield Therapy
Status: Completed | Type: Observational
Sponsor: MOA Health Science Foundation (Other)
Responsible Party: Principal Investigator, Kiyoshi Suzuki, President, MOA Health Science Foundation
Other Study IDs: MOA-004
Record Dates: First submitted 2019-06-17; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Pain; Depression, Anxiety; Dizziness; Signs and Symptoms
Keywords: biofield therapy; ethnic differences; Okada Purifying Therapy; effectiveness; safety
MeSH Terms: conditions — Pain; Depression; Anxiety Disorders; Dizziness; Signs and Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Okada Purifying Therapy — The practitioner raises his/her hand forward towards the recipient with the palm directed toward the recipient. The practitioner uses his/her hands alternately during the administration of Okada Purifying Therapy. The distance between the palm and the body is usually 1-2 feet, with each session typically lasting 30 to 60 minutes.

SUMMARY:
Participants from 14 different countries received a single session of biofield therapy (Okada Purifying Therapy) lasting 30 minutes or longer from the volunteer practitioners. Before and after the therapy, they reported the severity of physical pain, anxiety/depression, dizziness/palpitation, and overall symptoms. The team compared the effectiveness/safety of biofield therapy between countries and analyzed the factors associated with the outcomes.

DETAILED DESCRIPTION:
Participants aged 16 or older from 14 different countries (Japan, USA, Argentina, Brazil, Chile, Mexico, Peru, Taiwan, Thai, South Korea, Belgium, France, Portugal, and Spain) received a single session of biofield therapy (Okada Purifying Therapy) lasting 30 minutes or longer from the volunteer practitioners in their country of residence. Before and after the intervention, they reported each severity level of physical pain, anxiety/depression, dizziness/palpitation, and overall symptoms. The team compared the improvement/exacerbation rate of a single session of biofield therapy between the countries, and examined the adjusted odds ratio of the variables associated with the changes in each category of symptoms in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who agreed to receive a single session of biofield therapy for 30 minutes or longer from the volunteer investigators.
2. Individuals who were able to self-evaluate the change of their symptoms.
3. Individuals who were competent to answer the questionnaires.
4. Individuals who were aged 16 or older.

Exclusion Criteria:

* no specific exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants were recruited in various settings, including the workshop, the investigator's house, or the participant's home in 14 different countries.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2010-09-30 (Actual); Study Completion 2010-09-30 (Actual)

PRIMARY OUTCOMES:
improvement/exacerbation rate of symptoms after a single session of biofield therapy | Up to one year after all the data were collected.
  The Mann-Whitney test was conducted to compare the improvement/exacerbation rates between countries.
adjusted odds ratio of the factors associated with the changes in symptoms | Up to one year after all the data were collected.
  Logistic regression analyses

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Suzuki, MD, PhD, Study Chair — MOA Health Science Foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suzuki K, Uchida S, Kimura T, Tanaka H, Katamura H. International Cross-Sectional Study on the Effectiveness of Okada Purifying Therapy, a Biofield Therapy, for the Relief of Various Symptoms. J Altern Complement Med. 2020 Aug;26(8):708-720. doi: 10.1089/acm.2019.0264. Epub 2020 Jun 17. PMID 32551797